CLINICAL TRIAL: NCT03038542
Title: Quit4hlth: Enhancing Tobacco and Cancer Control Through Framed Text Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00044521
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Text Arm (Experimental)
  Interventions: Behavioral: Gain-framed text messages
- Standard Text Arm (Active Comparator)
  Interventions: Behavioral: Standard care text messages

INTERVENTIONS:
Behavioral: Gain-framed text messages
  Arms: Treatment Text Arm
Behavioral: Standard care text messages
  Arms: Standard Text Arm

SUMMARY:
This study evaluates a text messaging intervention through a smokers' quitline. Smokers will either receive 30 weeks of tailored, gain-framed text messages or 30 weeks of tailored, standard care text messages, both combined with standard quitline treatment. We hypothesize that the gain-framed text message intervention will increase cessation rates at 30 weeks as compared to standard care text messages.

ELIGIBILITY:
Inclusion Criteria:

* 1) call the Quitline requesting assistance with quitting smoking, 2) be 18+ years old, 3) speak English, 4) have a verified New York address, and 5) opt into the standard Quitline texting protocol.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
survey of smoking status | Week 30
  smoking or abstinent

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, PhD, Principal Investigator — Medical University of South Carolina